CLINICAL TRIAL: NCT06369116
Title: A Controlled, Observed Trial of Hepatitis C Self-Testing in the Hands of Untrained Lay Users
Brief Title: Trial of Hepatitis C Self-Testing in the Hands of Untrained Lay Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: bioLytical Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: CLS-017B; HSTAR012 (Other: HSTAR Programme); WRHI071 (Other: Ezintsha)
Record Dates: First submitted 2024-04-08; First posted 2024-04-16 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: Participants are recruited and enrolled to conduct INSTI HCV Self Test and then participate in the usability portion of the study.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Performance (Experimental): INSTI HCV Self Test devices are provided to the enrolled participants to conduct the self test using the provided instruction for use (IFU) as they are observed by a healthcare professional. The healthcare professional records observations while the participant is performing the self test and interpret the results. The trained healthcare professional is responsible for verifying the self-test result interpreted by the participant and further running another INSTI HCV Self-test to compare the results.
  Interventions: Device: INSTI HCV Self Test
- Usability and Label Comprehension (No Intervention): Participants are provided a usability and label comprehension questionnaire to score their experience with the INSTI HCV Self Test by referring to the provided Instruction For Use (IFU).

INTERVENTIONS:
Device: INSTI HCV Self Test — Each participant will be presented with a packaged self-test and asked to conduct self testing. The Trained Observer will only watch the participant process at a short distance and take notes on the process; at no point will the observer respond to questions or assist with the testing process - only to encourage the participant to try to figure out the process as best they can use the instruction sheet.
  The participant will then be permitted to perform the self-test and read their self test result. The observer is also going to observe the test result interpreted by the lay user and also themselves. After this step is complete, the Trained Observer will then perform fingerstick sample collection from lay user and run the sample on INSTI® HCV Self Test. The Trained Observer will then draw a venous whole blood sample from the participant for laboratory testing and final diagnosis will be given to the participant once laboratory results have been received.
  Arms: Performance

SUMMARY:
This is a controlled study intended to evaluate the usability, label comprehension and performance of the INSTI® HCV Self Test in the hands of untrained lay users using fingerstick blood, with instructions for use specifically designed for a lay person who has not used any hepatitis C rapid self test prior to the study and to assess "lay" users ability to comprehend key concepts and information provided on the outside of the pouch and in the accompanying Instructions for Use. Comprehension will be assessed without product familiarization (demonstration/training) by a healthcare professional.

DETAILED DESCRIPTION:
The HSTAR012 is a controlled study intended to evaluate the usability, label comprehension and performance of the INSTI® HCV Self Test in the hands of untrained lay users using fingerstick blood, with instructions for use specifically designed for a lay person who has not used any hepatitis C rapid self test prior to the study and to assess "lay" users ability to comprehend key concepts and information provided on the outside of the pouch and in the accompanying Instructions for Use. Comprehension will be assessed without product familiarization (demonstration/training) by a healthcare professional.

Specific critical and non-critical steps are identified from the self-test product's Instructions for Use. The untrained lay user is evaluated for process success or difficulty by a silent, non-interacting observer in the same room. Overall processes include self-test Usability (observation to determine if a participant performs all critical steps correctly), Interpretation of results (confirmation by staff to determine if participant interprets their test correctly), and labelling Comprehension (questionnaire to determine that the participant is aware of test limitations and what to do following the test result). The successful completion of steps will be evaluated as a percentage of the overall process, with all critical and non-critical errors identified and reported. All self-test results will be confirmed by testing with the same test by collecting additional fingerstick samples by a trained HCP (aka. Trained Observer). The level of agreement between the results of the investigated test (i.e., INSTI® HCV Self Test) obtained by a lay user and those obtained by a healthcare worker will be calculated.

Additionally, EDTA venous blood samples will be collected from each participant and sent to a laboratory to perform an enzyme immunoassay (EIA) using a state-of-the-art quality-assured assay (prequalified by WHO, CE-IVD or FDA approved). The sensitivity and specificity of the INSTI® HCV Self Test will be also calculated and the results from both tests conducted by the lay user and trained HCP compared to the results of the laboratory assay.

In the event of discrepant results between INSTI® HCV Self Test and the laboratory-based EIA assay, EDTA venous whole blood will be collected to perform HCV RNA assay to confirm active infection, study participants with positive results in HCV RNA test will be contacted and linked to care following local algorithms.

Study Aim

1. To evaluate the ability of untrained lay users to obtain an accurate test result using the INSTI® HCV Self Test.
2. To evaluate the untrained lay users' interaction with the device in terms of effectiveness and efficiency, i.e., successful/unsuccessful completion and difficulty of the critical steps as per the Instructions for Use.
3. To evaluate the performance (diagnostic sensitivity and specificity) of INSTI® HCV self-test by the lay user in comparison with laboratory confirmatory test.
4. To evaluate the performance (diagnostic sensitivity and specificity) of INSTI® HCV self-test by the healthcare professional in comparison with laboratory confirmatory test.
5. To evaluate the concordance of the results between the trained observer and the untrained lay user
6. To assess the ability of untrained lay users to correctly comprehend key messaging from device packaging and labelling, including the Instructions for Use.
7. To understand the experience and satisfaction of study participants with the overall self-testing process.
8. To assess whether or not the participants locate and read the information included in the IFU, know what the products are used for, and when it's appropriate/inappropriate to use the product.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Understand and sign the written informed Consent Form in English
* Have unknown HCV serology status, i.e., never tested for HCV or tested negative but the last testing was done at least 6 months before the enrolment date.
* Able to complete the required testing on the allocated testing day[s]
* Agree to provide accurate medical history, required specimens of finger prick blood samples for self-test devices, and up to 3.5ml of blood by venipuncture for laboratory testing.
* Able to speak and read English.

Exclusion Criteria:

* Do not meet all of the inclusion criteria.
* Are known HCV positive.
* Have received any experimental HCV vaccine.
* Have participated in any prior, or concurrent studies of self-testing including any blood based RDTs.
* A practicing medical healthcare professional (doctor, nurse or Counsellor that performs testing with RDTs)
* Any condition which, in the opinion of the facilitator, would make the participant unsuitable or unsafe for enrolment or could interfere with the completion of the assessment, consent form and questionnaire etc. or bias the outcome, i.e., being unable to see / read by forgetting to bring reading glasses, being intoxicated or acute sickness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1415 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Clinical sensitivity and specificity of INSTI HCV Self Test | 6 Months
  To evaluate the concordance between the results obtained by untrained lay users self-test to those results obtained by the HCP using another self-test device and lab-based confirmatory test and to ascertain the clinical sensitivity and specificity of the HCV Self-Test when compared to an approved state-of-the-art laboratory test.

SECONDARY OUTCOMES:
To assess the usability and label comprehension of the INSTI HCV Self Test | 1 month
  To assess the usability and label comprehension of the self-testing device and the ability of the participant to correctly comprehend the Instruction For Use of the self-test by observation of the self-testing procedure and documenting effectiveness and efficiency, i.e., successful / unsuccessful completion and difficulty of the critical steps as per the Instructions for Use. The label comprehension scoring spans from exceptionally satisfactory (score 5) to completely unsatisfactory (score 1).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Majam, Principal Investigator — Ezintsha, a division of Wits Health Consortium (Pty) Ltd
Locations (1):
- Ezintsha, a division of Wits Health Consortium (Pty) Ltd, Parktown, South Africa

IPD SHARING:
Plan to Share IPD: No